CLINICAL TRIAL: NCT04844320
Title: THE EFFECT OF FAST WEIGHT EFFICIENCY AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY ON THE COBB ANGLE IN MORBID OBESE PATIENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, MD. Anil Ergin, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR. ANIL ERGIN
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Obesity, Morbid; Back Pain; Scoliosis
Keywords: Morbid obesity; cobb angle; laparoscopic sleeve gastrectomy; scoliosis
MeSH Terms: conditions — Obesity, Morbid; Back Pain; Scoliosis

STUDY DESIGN:
Intervention Model Description: This study was designed to include 3 groups of 30 patients and a total of 90 patients. 90 patients who underwent laparoscopic sleeve gastrectomy will be divided into 3 groups according to their postoperative weight gain. The first group will include patients who have lost more than 50% EWL postoperative weight, the second group will include patients who have lost 50 to 25% EWL postoperative , and the third group will include patients who have lost less than 25% EWL postoperative.
  Patients in these 3 groups will be randomized on www.randomisor.org. In these 3 groups, cobb angle measurements will be made on the PA chest radiographs taken at the preoperative, postoperative 1st year and postoperative 2nd year controls. Patient satisfaction questionnaires will be conducted to compare pre- and postoperative complaints such as low back pain, back pain, and neck pain in all patients. The change in cobb angles will be determined according to the weight loss ratio (% EWL) of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- > 50 %EWL (Active Comparator): Postoperative weight loss in first year > 50 % EWL
  Interventions: Diagnostic Test: Cobb angle measurements
- 50 - 25 % EWL (Active Comparator): Postoperative weight loss in first year 25 - 50 % EWL
  Interventions: Diagnostic Test: Cobb angle measurements
- < 25 % EWL (Active Comparator): Postoperative weight loss in first year < 25 % EWL
  Interventions: Diagnostic Test: Cobb angle measurements

INTERVENTIONS:
Diagnostic Test: Cobb angle measurements — PA Chest x-rays will be taken in all patients in the preoperative, postoperative 1st year and 2nd year

SUMMARY:
Obesity has become an increasingly common health problem today. In this context, although many anatomical, physiological and metabolic problems arising from obesity in morbid obese patients are tried to be solved in daily practice, it has been proven that eliminating obesity is sufficient in the treatment of many diseases. When we look at the literature, it is known that morbid obesity causes deformation and excessive wear in most body joints. When morbid obesity disappears, it has been shown that the previously existing neck, waist, back and knee pains regress.

The aim of this study is to reveal the Cobb angle change in morbidly obese patients who achieved rapid weight loss after obesity surgery; To investigate the effect of weight loss on vertebral anatomy.

DETAILED DESCRIPTION:
90 morbidly obese patients who underwent Laparoscopic Sleeve Gastrectomy were included in the study. Cobb angle measurements were made by a radiologist included in the study from the PA chest radiographs of the operated patients in the preoperative period and in the first postoperative year, and they were recorded in a previously prepared database. In addition, in the preoperative period and postoperative first year evaluations of the patients; Patient satisfaction questionnaire in terms of low back pain, back pain, neck pain, and the value in% EWL of weight given after surgery were also recorded in the database.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18.
* Patients with a diagnosis of morbid obesity, body mass index> 40

Exclusion Criteria:

* Patients who have undergone previous vertebral surgery due to any disease
* Patients hospitalized for more than 10 days due to postoperative complications

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Cobb angle measurements | 2 years
  Cobb angle measurements will be made and recorded by an expert radiologist from the PA Chest X-ray.

SECONDARY OUTCOMES:
% EWL measurements | 2 years
  % EWL measurements will be made in all patients 1 and 2 years after laparoscopic sleeve gastrectomy
Patient satisfaction | 2 years
  All patients will be given a patient satisfaction questionnaire, which includes the complaints of low back pain, back pain and neck pain, and compares the postoperative and pre-operative processes.

CONTACTS AND LOCATIONS:
Locations (1):
- Anıl Ergin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No